CLINICAL TRIAL: NCT02781558
Title: A Phase 2, Multicenter, Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination (FDC) and Sofosbuvir/Velpatasvir FDC and Ribavirin in Subjects With Chronic Genotype 3 HCV Infection and Cirrhosis
Brief Title: Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination (FDC) and Sofosbuvir/Velpatasvir FDC and Ribavirin in Participants With Chronic Genotype 3 HCV Infection and Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-2097; 2016-000417-73 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SOF/VEL (Experimental): SOF/VEL FDC for 12 weeks
  Interventions: Drug: SOF/VEL
- SOF/VEL + RBV (Experimental): SOF/VEL FDC + RBV for 12 weeks
  Interventions: Drug: SOF/VEL; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: SOF/VEL + RBV

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) and SOF/VEL FDC and ribavirin (RBV) for 12 weeks in participants with chronic genotype 3 hepatitis C virus (HCV) infection and compensated cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* Individuals with chronic genotype 3 HCV infection and compensated cirrhosis
* Individuals with or without HIV-1 coinfection

Key Exclusion Criteria:

* History of clinically significant illness or any other medical disorder that may interfere with individual's treatment assessment or compliance with the protocol
* Co-infection with active hepatitis B virus
* Laboratory results outside the acceptable ranges at screening
* Pregnant or nursing female
* Chronic liver disease not caused by HCV

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (28):
- Spain (28):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital General Universitario De Alicante, Alicante
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Valle Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Servei de d'Aparell Digestiu Corporació Sanitària Parc Taulí, Barcelona
  - Reina Sofía University Hospital, Córdoba
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Puerta De Hierro Majadahonda, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen De La Arrixaca, Murcia
  - Hospital Universitario Central de asturias, Oviedo
  - Complexo Hospitalario Universitario de Montecelo, Pontevedra
  - Hospital Univ. NuestraSeñora Candelaria, Santa Cruz de Tenerife
  - Hospital de Valme, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario, Valencia
  - Hospital General Valencia, Valencia
  - La Fe Hospital, Valencia
  - Hospital Universitario Alvaro Cunqueiro, Vigo
  - Hospital Clinico Universitario, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Esteban R, Pineda JA, Calleja JL, Casado M, Rodriguez M, Turnes J, Morano Amado LE, Morillas RM, Forns X, Pascasio Acevedo JM, Andrade RJ, Rivero A, Carrion JA, Lens S, Riveiro-Barciela M, McNabb B, Zhang G, Camus G, Stamm LM, Brainard DM, Subramanian GM, Buti M. Efficacy of Sofosbuvir and Velpatasvir, With and Without Ribavirin, in Patients With Hepatitis C Virus Genotype 3 Infection and Cirrhosis. Gastroenterology. 2018 Oct;155(4):1120-1127.e4. doi: 10.1053/j.gastro.2018.06.042. Epub 2018 Jun 27. PMID 29958855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Spain. The first participant was screened on 29 July 2016. The last study visit occurred on 27 October 2017.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) 400/100 mg fixed-dose combination (FDC) tablet once daily for 12 weeks
- SOF/VEL + RBV: SOF/VEL 400/100 mg FDC tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL | SOF/VEL + RBV
Started | 101 | 103
Completed | 98 | 101
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of any study drug
Groups:
- SOF/VEL: SOF/VEL 400/100 mg FDC tablet once daily for 12 weeks
- SOF/VEL + RBV: SOF/VEL 400/100 mg FDC tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL | SOF/VEL + RBV | Total
Number analyzed (Participants) | 101 | 103 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (7.3) | 51 (7.6) | 51 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 16 | 42
  Male | 75 | 87 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 84 | 95 | 179
  Asian | 17 | 8 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 92 | 93 | 185
IL28B [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 64 | 53 | 117
    Non-CC | 36 | 50 | 86
    Missing | 1 | 0 | 1
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.64) | 6.3 (0.56) | 6.2 (0.60)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 32 | 24 | 56
  ≥ 800,000 IU/mL | 69 | 79 | 148

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Cessation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all randomized participants who took at least 1 dose of any study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL + RBV: SOF/VEL 400/100 mg FDC tablet once daily RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 101 | 103
percentage of participants | 91.1 [83.8 to 95.8] | 96.1 [90.4 to 98.9]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug (Which Included SOF/VEL and RBV) Due to Any Adverse Event
Time Frame: Posttreatment Week 12
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 101 | 103
percentage of participants | 1.0 | 1.9

3. Secondary Outcome: Percentage of Participants Who Attain Sustained Virologic Response at 4 Weeks After Cessation of the Study Treatment Regimen (SVR4)
Description: SVR4 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 101 | 103
percentage of participants | 93.1 [86.2 to 97.2] | 97.1 [91.7 to 99.4]

4. Secondary Outcome: Percentage of Participants Who Have HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 103
percentage of participants | 51.0 [40.8 to 61.1] | 44.7 [34.9 to 54.8]

5. Secondary Outcome: Percentage of Participants Who Have HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 103
percentage of participants | 85.0 [76.5 to 91.4] | 90.3 [82.9 to 95.2]

6. Secondary Outcome: Percentage of Participants Who Have HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 102
percentage of participants | 99.0 [94.6 to 100.0] | 100.0 [96.4 to 100.0]

7. Secondary Outcome: Percentage of Participants Who Have HCV RNA < LLOQ at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 101
percentage of participants | 99.0 [94.6 to 100.0] | 100.0 [96.4 to 100.0]

8. Secondary Outcome: HCV RNA at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 97 | 102
log10 IU/mL | 1.52 (0.513) | 1.47 (0.413)

9. Secondary Outcome: HCV RNA at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 103
log10 IU/mL | 1.22 (0.257) | 1.19 (0.152)

10. Secondary Outcome: HCV RNA at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 102
log10 IU/mL | 1.15 (0.040) | 1.15 (0.000)

11. Secondary Outcome: HCV RNA at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 101
log10 IU/mL | 1.15 (0.018) | 1.15 (0.000)

12. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 97 | 102
log10 IU/mL | -4.67 (0.627) | -4.80 (0.580)

13. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 103
log10 IU/mL | -4.96 (0.641) | -5.09 (0.559)

14. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 102
log10 IU/mL | -5.04 (0.638) | -5.13 (0.565)

15. Secondary Outcome: Change From Baseline in HCV RNA at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 100 | 101
log10 IU/mL | -5.04 (0.640) | -5.13 (0.568)

16. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ on 2 consecutive measurements while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement
Time Frame: Up to Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 101 | 103
percentage of participants | 5.9 | 1.9

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL | SOF/VEL + RBV
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/103
Serious Adverse Events (participants affected / at risk) | 4/101 | 2/103
Other Adverse Events (participants affected / at risk) | 24/101 | 55/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=101) | SOF/VEL + RBV (N=103)
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Accident at work (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=101) | SOF/VEL + RBV (N=103)
Nausea (Gastrointestinal disorders) | 2 | 6
Asthenia (General disorders) | 12 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Headache (Nervous system disorders) | 8 | 25
Insomnia (Psychiatric disorders) | 1 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT02781558/Prot_000.pdf
  • Study Protocol: Protocol Amendment 1 (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT02781558/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT02781558/SAP_002.pdf